CLINICAL TRIAL: NCT02642822
Title: The Epidemiologic Study of Human Cytomegalovirus （CMV）in Female Students of Xiamen University
Brief Title: The Epidemiologic Study of Human Cytomegalovirus（CMV） in Female Students of Xiamen University
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, vice dean of School of Public Health, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: CMV-EPI-002
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2015-12

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, 100 female students aged 18 to 30 years old in Xiamen University will be enrolled. On the first visit, blood, saliva and urine samples of all participants will be collected. Then saliva and urine samples will be collected at two-week interval until 6 months. Serum samples will be tested the PP150-IgG titer. Saliva and urine samples will be used to test CMV DNA by PCR. The primary purpose of this study is to identify the relationship between baseline PP150-IgG titer and CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* female students of Xiamen University

Exclusion Criteria:

* students who have the serious diseases

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 female students aged 18 to 30 years old will be recruited from Xiamen University.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
rate of active CMV infection in different PP150-IgG titer | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health of Xiamen University, Xiamen, Fujian, China